CLINICAL TRIAL: NCT06743022
Title: Evaluation of the Reproducibility of the Automated Measurement of the Extent of Interstitial Lung Disease on Chest CT
Brief Title: Evaluation of the Reproducibility of the Automated Measurement of the Extent of ILD on Chest CT
Acronym: REPRO-PID
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP240783; 2024-A01384-43 (Other: France : Ministry of Health)
Record Dates: First submitted 2024-12-16; First posted 2024-12-19 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Interstitial Lung Disease
Keywords: Lung Diseases; Interstitial Lung Disease; Multidetector Computed Tomography; Deep Learning
MeSH Terms: conditions — Lung Diseases, Interstitial; Lung Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Patients with interstitial lung disease (Experimental)
  Interventions: Diagnostic Test: Chest CT

INTERVENTIONS:
Diagnostic Test: Chest CT — Repeated chest CT for automated ILD quantification

SUMMARY:
In interstitial lung disease (ILD), the extent of ILD on chest computed tomography (CT) is recognized as an important prognostic factor. Automated tools are now available to quantify ILD, but there is a lack of data on the reproducibility of this measurement and therefore its accuracy.

Therefore, the purpose of this study is to evaluate the variability of automated ILD quantification on chest CT. Reproducibility will be assessed by repeating chest CT scans and using different tools to measure the extent of disease.

DETAILED DESCRIPTION:
In interstitial lung disease (ILD), the extent of ILD on chest computed tomography (CT) is recognized as an important prognostic factor. In recent years, several tools based on texture analysis or deep learning methods have been developed to provide rapid and accurate automated quantification of ILD extent.

An advantage of automated scoring methods is that they theoretically offer perfect repeatability of measurement. However, this is only true if the measurement is repeated on the same images. Several parameters can alter the appearance of the lungs on scanner images, such as the degree of inspiration or the reconstruction kernel used to reconstruct the images. There is a lack of data on the reproducibility of the whole process of automated ILD quantification and therefore its accuracy.

Therefore, the purpose of this study is to evaluate the variability of automated ILD quantification on chest CT.

Reproducibility will be assessed by repeating chest CT scans and using different tools to measure the extent of disease in patients with ILD from 2 institutions. Chest CT will be repeated the same day. This will allow assessment of the variability of automated measurement of ILD extent between 2 CT scans performed on the same day and when using different software. It will also allow to assess the variability of lung volume between the 2 CT scans and the effect of disease (idiopathic pulmonary fibrosis or connective tissue disease-related ILD) on the reproducibility of ILD quantification.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Known interstitial lung disease as part of idiopathic pulmonary fibrosis or connective tissue disease
* Followed in one of the participating hospitals
* Requiring a chest CT as part of a scheduled assessment
* Affiliated to a French national social security
* Informed consent

Exclusion Criteria:

* Acute exacerbation of ILD
* Pregnancy
* Inability to hold an apnea for 10 seconds
* Patients in the exclusion period after a previous research
* Need for additional procubitus or expiratory images

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-06-24 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Automated Interstitial Lung Disease (ILD) quantification | Day of inclusion
  Reproducibility of ILD quantification on chest CT (as a percentage of lung volume) between two successive scan acquisitions.

SECONDARY OUTCOMES:
Automated Interstitial Lung Disease (ILD) quantification | Day of inclusion
  Reproducibility of disease extent measured with different software on the same acquisition
Lung volume | Day of inclusion
  Reproducibility of total lung volume measured on the scanner between two successive acquisitions
Automated Interstitial Lung Disease (ILD) quantification | Day of inclusion
  Reproducibility of disease extension between the two scan acquisitions depending on the disease (idiopathic pulmonary fibrosis or PID secondary to connective tissue disease).

CONTACTS AND LOCATIONS:
Overall Officials: Guillaume CHASSAGNON, MD, PhD, Principal Investigator — Cochin Hospital - AP-HP
Locations (6):
- France (6):
  - APHP - Bichat hospital - Radiology, Paris, IDF
  - APHP - Bichat hospital - Rheumatology, Paris, IDF
  - APHP - Cochin Hospital - Internal medicine, Paris, IDF
  - APHP - Cochin Hospital - Pneumology, Paris, IDF
  - APHP - Cochin Hospital - Radiology, Paris, IDF
  - APHP - Bichat Hospital - Pneumology, Paris, IDF

IPD SHARING:
Plan to Share IPD: No